CLINICAL TRIAL: NCT01163539
Title: Cyberknife Radiosurgery and Quality of Life
Status: Terminated | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: SPN0002; SU-07092010-6499 (Other: Stanford University)
Record Dates: First submitted 2010-07-14; First posted 2010-07-15 (Estimated); Last update posted 2016-07-01 (Estimated); Status verified 2016-06

CONDITIONS: Bone Cancer; Central Nervous System Cancer
MeSH Terms: conditions — Bone Neoplasms; Central Nervous System Neoplasms

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to look at pain control and QOL improvement after treatment with CK Radiosurgery for spinal metastases.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a spinal metastasis who will be treated with Cyberknife radiosurgery.
* There are no age or gender restrictions.
* There are no life expectancy restrictions.
* Karnofsky Performance Status greater than 40.
* Negative pregnancy test or clinically assessed as not pregnant.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients with benign tumors will not be included (neurofibromas, schwannomas, etc.)
* Other investigational medications or treatments will be noted, but will not preclude inclusion.
* Pregnant or nursing patients will be not be included in the study due to radiation exposure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient must have cancer metastases to the spine. They may have had previous surgical or not surgical treatments. Benign tumors will not be assessed.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2010-07; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Daniel Chang, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States